CLINICAL TRIAL: NCT02364544
Title: The Improving Care and Reducing Cost (ICRC) Program
Brief Title: Improving Care and Reducing Cost Study
Acronym: ICRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: University of Pittsburgh (Other); Boston University (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John Kane, Senior Vice President, Behavioral Health Services, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICRC
Record Dates: First submitted 2015-01-30; First posted 2015-02-18 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychosis NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Health Technology Program (Other): The components of the treatment model include: 1) Prescriber Decision Assistant (PDA) 2) relapse prevention plan, 3) the daily support website 4) FOCUS, an interactive smart phone text-messaging application 5) a web-based, cognitive-behavioral therapy (CBT) program
  All patients will be provided with pharmacological treatment (PDA), brief in-person relapse prevention counseling, and an Android mobile phone. The other program components will be provided to patients using a shared decision-making approach to assess need and preference.
  Interventions: Behavioral: Relapse Prevention Plan; Behavioral: Daily Support Website; Behavioral: Computer CBT for voices and paranoia; Behavioral: FOCUS; Other: Prescriber Decision Assistant

INTERVENTIONS:
Behavioral: Relapse Prevention Plan — brief, in-person, relapse prevention counseling with supplemental web-based learning modules,
Behavioral: Daily Support Website — web-based program for patients and families that provides psychoeducation about schizophrenia and its treatments to improve knowledge, increase problem-solving skills and offer social support through the use of web-based therapist facilitated sessions
Behavioral: Computer CBT for voices and paranoia — A ten-session CBT programs, one to address voices and the other for paranoia. The web-based programs incorporate the essential elements of CBT for psychosis such as normalizing behavior and offering behavioral coping strategies
Behavioral: FOCUS — an interactive smart phone text-messaging application to support medication adherence, facilitate coping with symptoms and improve daily functioning in individuals with schizophrenia
Other: Prescriber Decision Assistant — is a web-based prescriber decision support system that includes a brief patient-completed assessment describing symptoms and adverse events which prompts the prescriber to conduct a detailed clinical assessment. Embedded in the program are decision supports for medication choices based on best evidence-based practices regarding symptoms, side effects, information from laboratory tests and history of prior treatment response

SUMMARY:
The goal of the Improving Care and Reducing Cost (ICRC) Program, is to improve disease management and the overall process of care in treating the chronic illness schizophrenia in order to reduce ER visits and hospital days while providing better care, better health and increased patient satisfaction. This will be done by fostering innovation in the use of technology and by training and deploying a new cadre of personnel in the behavioral health field: Mental Health/Health Technology (MH/HT) Case Managers.

DETAILED DESCRIPTION:
The goal of the Improving Care and Reducing Cost (ICRC) Program, is to improve disease management and the overall process of care in treating the chronic illness schizophrenia in order to reduce ER visits and hospital days while providing better care, better health and increased patient satisfaction. This will be done by fostering innovation in the use of technology and by training and deploying a new cadre of personnel in the behavioral health field: Mental Health/Health Technology (MH/HT) Case Managers. The specific treatments we propose to use are evidence based, but their dissemination has been limited because of lack of trained personnel and cost. The model we propose, the Health Technology Program (HTP), will address these problems through use of the web and mobile phone based training and interventions.

The components of the HTP program that are being tested in the pilot program include: 1) evidence-based pharmacological treatment facilitated by a web-based prescriber decision support system-Prescriber Decision Assistant (PDA) 2) brief, in-person, relapse prevention counseling with supplemental web-based learning modules, 3) a daily support website that offers web- and phone-based resources to support persons with schizophrenia and their family members or others. The resources include a patient and family Psycho-Education Treatment program, which includes electronic peer groups facilitated by mental health professionals, providing medication reminders via web and phone, and conducting monitoring of early warning signs of relapse via web and phone 4) an interactive smart phone text-messaging application to support medication adherence, facilitate coping with symptoms and improve daily functioning in individuals with schizophrenia 5) a web-based, self-administered cognitive-behavioral therapy (CBT) program for the management of hallucinations. All patients will be provided with pharmacological treatment (PDA), brief in-person relapse prevention counseling, and an Android mobile phone. The other program components will be provided to patients using a shared decision-making approach to assess need and preference.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 60, (patients age 51-60 require review from the coordinating site)

  * Clinical diagnosis of:

    * schizophrenia
    * schizoaffective disorder
    * psychosis NOS
  * Has had two or more inpatient hospitalizations for treatment of a psychotic disorder
  * Currently in the hospital or up to 30 days of inpatient hospitalization for a psychotic disorder

    o If patients are sent to a partial, or day hospital following an inpatient hospitalization, the 30 day window begins at the time of discharge from the day or partial hospital
  * Any ethnicity
  * Ability to participate in research assessments in English
  * Ability to provide fully informed consent

Exclusion Criteria:

* • Individuals who cannot understand what research participation entails, or correctly answer the questions about research participation that are part of the Study Information Review and provide fully informed consent will be excluded

  * More than 30 days since discharge from a psychiatric hospitalization
  * Any other serious medical condition that in the opinion of the investigator would seriously impair functioning making the patient unsuitable for the trial
  * Patients who would likely find it burdensome and/or have difficulty sustaining the use of a laptop computer and /or smart phone due to issues of security, consistent connectivity or other factors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 461 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total Number of Hospitalization and Emergency Room Visits | Baseline, Month 1, Month2, Month 3, Month4, Month 5, and Month 6
  Captures the number of hospital and ER visits each month

SECONDARY OUTCOMES:
Service Utilization Resource Form | Baseline, month 3, month 6
  Captures services received in the last 30 days
Change from Baseline Heinrich's Quality of Life Scale | Baseline and month 6

CONTACTS AND LOCATIONS:
Overall Officials: John Kane, Principal Investigator — Northwell Health
Locations (8):
- United States (8):
  - Henderson Mental Health Center, Fort Lauderdale, Florida
  - Community Mental Health Center, Inc., Lawrenceburg, Indiana
  - Cherry Street, Grand Rapids, Michigan
  - UMKC School of Pharmacy, Kansas City, Missouri
  - Burrell Behavioral Health, Springfield, Missouri
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - University of New Mexico Department of Psychiatry UNM Health Sciences Center, Albuquerque, New Mexico
  - PeaceHealth Oregon/Lane County Behavioral Health Services, Eugene, Oregon